CLINICAL TRIAL: NCT03263611
Title: A Phase 1b, Multicenter, Double-blind, Randomized, Placebo-controlled, Single Ascending-Dose, Clinical Study Evaluating the Safety, Tolerability and Exploratory Efficacy of a Targeted Single Injection of an Intradiscal Nuclear Factor-κB Decoy Oligodeoxynucleotide (AMG0103) in Subjects With Chronic Discogenic Lumbar Back Pain
Brief Title: AMG0103 in Subjects With Chronic Discogenic Lumbar Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnGes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMG0103-US-01
Record Dates: First submitted 2017-08-16; First posted 2017-08-28 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Degenerative Disc Disease
Keywords: disc degeneration; Intervertebral disc; discogenic pain; chronic discogenic lumbar back pain
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- placebo (Placebo Comparator): subject will receive single intradiscal injection of placebo
  Interventions: Drug: Placebo
- AMG0103 low dose (Experimental): subject will receive single intradiscal injection of AMG0103 low dose
  Interventions: Drug: AMG0103
- AMG0103 middle dose (Experimental): subject will receive single intradiscal injection of AMG0103 middle dose
  Interventions: Drug: AMG0103
- AMG0103 high dose (Experimental): subject will receive single intradiscal injection of AMG0103 high dose
  Interventions: Drug: AMG0103

INTERVENTIONS:
Drug: Placebo — single intradiscal injection
  Arms: placebo
Drug: AMG0103 — single intradiscal injection
  Arms: AMG0103 high dose; AMG0103 low dose; AMG0103 middle dose

SUMMARY:
This clinical trial evaluate the safety, tolerability and exploratory efficacy of targeted single injection of AMG0103 in subject with chronic discogenic lumbar back pain

DETAILED DESCRIPTION:
This is a Phase 1b, multicenter, double-blind, single ascending dose study designed to evaluate the safety of AMG0103 in adult male and female subjects with chronic discogenic lumbar back pain.

This protocol anticipates that 8 subjects with symptomatic single level discogenic pain will be enrolled in each of up to 3 dose-escalation cohorts. Subjects in each cohort will receive AMG0103 or Placebo as a targeted, single, intradiscal injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 75 years of age, inclusive, and skeletally mature, in the opinion of the investigator.
2. Has provided written informed consent before undergoing any study-specific procedures.
3. Has chronic low back pain for at least 6 months, where back pain is greater than leg pain.
4. Has separate low back pain and leg pain VAS scores within the following parameters:

   1. Average low back pain VAS score of at least 40 mm and less than 90 mm on a 100 mm visual analog scale.
   2. Average leg pain VAS score that is less than or equal to 50% of the average low back pain VAS score above, where leg pain VAS scores are measured on a 100 mm visual analog scale.
5. Has had inadequate response to conservative medical care over a period of at least 3 months.
6. Diagnosis of painful degenerative disc disease at one lumbar level from L1 to S1 confirmed by subject history and radiographic studies (eg, MRI, x-rays). Radiographic studies must demonstrate the following:

   1. A Pfirrmann score of 3 or 4 on MRI in just a single disc between L1 and S1
   2. With or without contained disc herniations of <3 mm protrusion with no radiographic evidence of neurologic compression
   3. Disc height loss of the symptomatic disc is less than 50% of the adjacent discs
   4. All discs other than the index disc must have a Pfirrman score of less than 3
   5. No spondylolisthesis or instability on flexion/extension views of more than 1-2 mm
   6. No evidence of sacroiliac, or extra-spinal, pathology that could account for lumbar back pain
   7. No more fluid in, or widening of, the facet joints around the symptomatic disc than is seen on the other facet joints of "normal" levels
7. Has a Body Mass Index (BMI) between 15.0 and 35.0 kg/m2 at the screening visit.
8. Oswestry Disability Index score of at least 30 and not more than 90 on the 100 point questionnaire.
9. Willing and able to comply with all protocol requirements.
10. Females of childbearing potential must agree to use highly effective methods of contraception during heterosexual intercourse from the date they sign the ICF until 1 year after the single dose of study drug is administered.
11. Male subjects must agree that, if their partner is of childbearing potential, they and the partner will use an appropriate method of contraception as defined above.

Exclusion Criteria:

1. Has any prior or current medical condition (eg, an active systemic infection), including known bleeding disorders that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all study requirements.
2. Has any clinically significant finding on a screening evaluation that in the judgment of the Investigator would preclude safe study completion.
3. Liver function tests >1.5 the upper limit of normal (ULN) for alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST)
4. Serum creatinine >1.5 ULN at screening
5. Blood pressure >160/110 mm Hg recorded on 3 readings at screening and/or resting pulse >120 beats/min at screening
6. Body temperature ≥101°F on day of planned injection
7. Has a co-morbid medical condition of the spine or the upper extremities that may affect neurological and/or pain assessments as specified in the protocol, including spinal fusion, spondylolysis and spondylolisthesis.
8. Has evidence of hip pathology based on clinical history, physical exam and/or radiographic imaging that could be the source of lumbar back pain.
9. Has a history of an endocrine or metabolic disorder that affects the spine (eg, Paget's disease).
10. Has a compressive pathology due to stenosis or frankly herniated disc or sequestered discs.
11. Has symptomatic involvement of more than one lumbar disc, in the opinion of the investigator.
12. Has an intact disc bulge/protrusion or focal herniation at the symptomatic level >3 mm, the presence of disc extrusion or sequestration, or a complete annular tear.
13. Has lumbar intervertebral foraminal stenosis at the symptomatic level resulting in clinically significant spinal nerve root compression, in the opinion of the investigator.
14. Has undergone a previous surgery at the symptomatic disc, or has plans to do so within 6 months of receiving the dose of AMG0103, that has altered the structure of the target disc level, or is likely to do so (eg, laminectomy, foraminotomy, fusion, intradiscal electrothermal therapy, intradiscal radiofrequency, thermocoagulation).
15. Has had any lumbar intradiscal injection procedure (eg, injection of corticosteroids, methylene blue, dextrose, or glucosamine and chondroitin sulfate). Discography may be performed, but must be done at least 3 weeks (or more) prior to the injection procedure in this study.
16. Has had any epidural steroid injection(s) within 3 months prior to study treatment.
17. Is a female who is pregnant, planning to become pregnant, or lactating.
18. Has a PT(INR) and/or aPTT lab result outside of the reference range, or within the last 30 days taken, or is currently on, an anticoagulant therapy (e.g., Warfarin) for the purpose of treating or preventing blood clots.
19. Has ferromagnetic implants that would disallow MRI of the symptomatic disc.
20. Is involved in current or pending spinal litigation where permanent disability benefits are being sought.
21. Has a physical or mental condition (eg, senile dementia, Alzheimer's disease) that would interfere with Subject self-assessment of function, pain or quality of life.
22. Has a positive screen for Hepatitis B Surface Antigen, Hepatitis C antibodies, or human immunodeficiency virus (HIV) by antibodies or nucleic acid test.
23. Is an immediate family member (by birth) of any other subject participating in this study.
24. Has a history of cancer that does NOT have documentation to support a complete and curative treatment.
25. Has participated within the previous 3 months in an interventional clinical study or is concurrently enrolled in any non-interventional research of any type judged to be scientifically or medically incompatible with this study.
26. Is transient or has been treated in the 6 months prior to providing informed consent for alcohol and/or drug abuse in an inpatient substance abuse program.
27. Is currently incarcerated (a prisoner).
28. Is an Investigator-site employee or immediate family (defined as a spouse, parent, child, or sibling, whether biological or legally adopted) of an Investigator-site employee.
29. Is a Sponsor employee (permanent, temporary contract worker, or designee responsible for the conduct of the study) or immediate family (defined as a spouse, parent, child, or sibling, whether biological or legally adopted) of a Sponsor employee.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Safety: treatment-emergent adverse events (AEs) | 6 months
Safety: data from 12-lead electrocardiograms | 6 months
Safety: data from clinical laboratory evaluations (hematology, serum chemistry, coagulation, inflammation and immunology) | 6 months

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) for pain | 6 months
Oswestry Disability Index to assess Activity of Daily Living | 6 months
Roland Morris Disability Questionnaire to assess Activity of Daily Living | 6 months
Patient Global Impression of Change pain self-assessment scale to assess Quality of Life | 6 months
SF-36 to assess Quality of Life | 6 months
Disc space height by X-ray | 6 months
Pfirrmann Score by MRI | 6 months
PK of AMG0103: Cmax | 1 month
  Maximum plasma concentration estimate for a single injection of AMG0103
PK of AMG0103: Tmax | 1 month
  Time to maximum plasma concentration estimate for a single injection of AMG0103
PK of AMG0103: AUC | 1 month
  Area under the plasma-concentration time curve (AUC) estimate for a single injection of AMG0103
Amount of AMG0103 excreted into urine | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: AnGes, Inc. Clinical Development, Study Director — AnGes, Inc.
Locations (6):
- United States (6):
  - Keck Medicine of USC, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Spine Institute of San Diego, San Diego, California
  - Florida Medical Pain Management, St. Petersburg, Florida
  - Florida Medical Relief, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Kato K, Akeda K, Miyazaki S, Yamada J, Muehleman C, Miyamoto K, Asanuma YA, Asanuma K, Fujiwara T, Lenz ME, Nakazawa T, An H, Masuda K. NF-kB decoy oligodeoxynucleotide preserves disc height in a rabbit anular-puncture model and reduces pain induction in a rat xenograft-radiculopathy model. Eur Cell Mater. 2021 Jul 20;42:90-109. doi: 10.22203/eCM.v042a07. PMID 34284523